CLINICAL TRIAL: NCT02983071
Title: Phase 1/2 Safety, Pharmacokinetic, and Antitumor Activity Study of G1T38 in Combination With Fulvestrant in Patients With Hormone Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer After Endocrine Failure
Brief Title: G1T38, a CDK 4/6 Inhibitor, in Combination With Fulvestrant in Hormone Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G1T38-02; 2016-001485-29 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Ductal, Breast; Breast Cancer; Breast Neoplasm
Keywords: Breast Cancer; CDK 4/6 Inhibitor; HER2-Negative; HR-Positive; HR+; HER2-; HER2 -ve; HER2 +ve
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once-Daily G1T38 Dosing (Experimental): G1T38 (lerociclib) orally (once daily) in combination with fulvestrant.
  Interventions: Drug: G1T38; Drug: Fulvestrant
- Twice-Daily G1T38 Dosing (Experimental): G1T38 (lerociclib) orally (twice daily) in combination with fulvestrant.
  Interventions: Drug: G1T38; Drug: Fulvestrant

INTERVENTIONS:
Drug: G1T38
  Other Names: lerociclib
Drug: Fulvestrant
  Other Names: Faslodex

SUMMARY:
This is a study to investigate the potential clinical benefit of G1T38 as an oral therapy in combination with fulvestrant in patients with hormone receptor-positive, HER2-negative metastatic breast cancer.

The study is an open-label design, consists of 2 parts: dose-finding portion (Part 1), and expansion portion (Part 2). Both parts include 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase begins on the day of first dose with study treatment and completes at the Post-Treatment Visit. Approximately, 102 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HR-positive, HER2-negative breast cancer, not amenable to curative therapy
* Pre- or perimenopausal women can be enrolled if amenable to be treated with goserelin
* Patients must satisfy 1 of the following criteria for prior therapy:

  * Progressed during treatment or within 12 months of completion of adjuvant therapy with an aromatase inhibitor or tamoxifen
  * Progressed during treatment or within 2 months after the end of prior aromatase inhibitor therapy for advanced/metastatic breast cancer, or prior endocrine therapy for advanced/metastatic breast cancer
  * Received ≤ 2 chemotherapy regimens (Part 1) or ≤ 1 chemotherapy regimen (Part 2) for advanced/metastatic disease
* For Part 1, evaluable or measurable disease (bone only disease eligible for Part 1 only)
* For Part 2, measurable disease as defined by RECIST, Version 1.1
* ECOG performance status 0 to 1
* Adequate organ function

Exclusion Criteria:

* For Part 1, prior treatment with fulvestrant
* For Part 2, prior treatment with any CDK inhibitor or fulvestrant
* Active uncontrolled/symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease
* Chemotherapy within 21 days of first G1T38 dose
* Investigational drug within 28 days of first G1T38 dose
* Concurrent radiotherapy, radiotherapy within 14 days of first G1T38 dose, previous radiotherapy to the target lesion sites, or prior radiotherapy to > 25% of bone marrow
* Prior hematopoietic stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2017-01; Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Week 1 Day 1-Week 5 Day 1
Recommended Phase 2 dose | 14 months
Recommended Phase 2 dose interval | 14 months
  Twice-Daily or Once-Daily dosing
Number of Treatment Related Adverse Event, including Abnormal Laboratory Events | 36 months
  All AEs, including clinical laboratory, vitals signs, physical examinations and ECGs will be analyzed in all patients receiving study drug from the signing of the informed consent until 30 days after the last dose of study medication up to 36 months

SECONDARY OUTCOMES:
Tumor response based on RECIST, Version 1.1 | 30 months
Pharmacokinetics of G1T38, Fulvestrant, and Goserelin: Maximum Plasma Concentration (Cmax) | Week 1 Day 1-Week 9 Day 1
Pharmacokinetics of G1T38, Fulvestrant, and Goserelin: Area under Curve - plasma concentration (AUC) | Week 1 Day 1-Week 9 Day 1
Pharmacokinetics of G1T38, Fulvestrant, and Goserelin: Plasma: terminal half life (T1/2) | Week 1 Day 1-Week 9 Day 1
Pharmacokinetics of G1T38, Fulvestrant, and Goserelin: Plasma - Volume of distribution | Week 1 Day 1-Week 9 Day 1
Progression free survival (PFS) | 36 months
Overall survival (OS) | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (8):
- Bulgaria (2):
  - MHAT for Womens Health - Nadezhda OOD, Sofia
  - Special Hospital For Active Treatment In Oncology, Sofia
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- The Institute of Oncology, Chisinau, Moldova
- United Kingdom (4):
  - Cambridge University, Cambridge
  - University College London Hospital (UCLH), London
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation, Manchester